CLINICAL TRIAL: NCT07080853
Title: Efficacy of a Novel Exercise + Overdressing Protocol to Induce Targeted Heat Stress in Temperate Environments (Acute XO-Study)
Brief Title: Acute Exercise With Overdressing
Acronym: Acute-XO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Army Research Institute of Environmental Medicine (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 23-14
Record Dates: First submitted 2025-07-02; First posted 2025-07-23 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Heat Stress, Exertional; Heat Acclimation and Thermotolerance
Keywords: Heat acclimation; Overdressing
MeSH Terms: conditions — Heat Stress Disorders | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise with Overdressing (Experimental): Exercise with overdressing clothing ensemble
  Interventions: Other: Exercise with Overdressing
- Control Exercise (Active Comparator): Exercise with normal attire
  Interventions: Other: Control Exercise

INTERVENTIONS:
Other: Exercise with Overdressing — Run for 30 minutes followed by walk for 60 minutes in a temperate (gym-like environment) wearing overdressing ensemble.
  Arms: Exercise with Overdressing
Other: Control Exercise — Run for 30 minutes followed by walk for 60 minutes in a temperate (gym-like environment) wearing control clothing ensemble.
  Arms: Control Exercise

SUMMARY:
The purpose of this study is to determine if exercise with extra clothing in a gym-like environment can increase body temperatures appropriately to help people adapt to the heat.

DETAILED DESCRIPTION:
The purpose of the present study is to examine the influence of a novel 90-minute exercise + overdressing protocol on thermal responses in comparison to matched exercise in standard PT clothing. Sixteen healthy and fit adults (8 men and 8 women) will complete two 90-minute exercise sessions (randomized order) in a temperate environment (~20°C, ~50% relative humidity, and ~1 mph air velocity) involving a 30-minute run immediately followed by a 60-minute walk. Participants will wear standard physical training (PT) clothing (shorts, t-shirt) during one session and an overdressing ensemble in the other. The investigators hypothesize that 1) exercise + overdressing will elevate core temperature to between 38.3°C and 39.3°C for at least 45 minutes; and 2) elevations in core temperature, skin temperature, heart rate, and sweat rate will be substantially larger than observed with 90 minutes of matched exercise in standard PT clothing.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 18-45
* Females must be premenopausal
* Body mass index 18.5-30.0 kg m-2
* In good health as determined by the Office of Medical Support & Oversight (OMSO) General Medical Clearance
* Performs aerobic exercise at least 2 times per week and capable of running 2 miles in under 16:00 (8 minute mile pace)
* Willing to abstain from exercise and alcoholic beverages for 24 hours before each study visit.
* Willing to abstain from caffeine for 12 hours prior to all study visits.
* Willing to abstain from food for 2 hours prior to all study visits.
* Willing to abstain from nicotine/tobacco for at least 8 hours prior to all study visits.
* Have supervisor approval if permanent party military or a federal employee at U.S. Army Natick Soldier System Center

Exclusion Criteria:

* Females who are pregnant or planning to become pregnant during the study
* Taking dietary supplements, prescriptions, or over the counter medication, other than a contraceptive (unless approved by OMSO & PI)
* Abnormal blood count during OMSO medical screening (For example: hemoglobin (Hb) outside of the typical normal values reported by LabCorp in accordance with OMSO (Normal [Hb] Males = 12.6-17.7 g/dL; Females = 11.1-15.9 g/dL) or hematocrit (Hct) outside of the normal ranges (Normal Hct Males = 37.5-51.0%; Females = 34.0-46.6%) levels, presence of abnormal blood chemicals (hemoglobin S or sickle cell traits)
* Any history of pulmonary or cardiovascular disease
* Any history of asthma
* Current or recent respiratory tract or sinus infections (< 1 month prior)
* History of heat intolerance or orthostatic intolerance
* Diagnosed and/or treated for fluid/electrolyte imbalance within the last 30 days
* History of obstructive disease of the gastrointestinal tract including (but not limited to) diverticulosis, diverticulitis and inflammatory bowel disease, peptic ulcer disease, Crohn's disease, ulcerative colitis.
* Scheduled MRI during testing
* Allergies to adhesives (e.g., medical tape).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2023-06-22 (Actual); Primary Completion 2025-04-28 (Actual); Study Completion 2025-04-28 (Actual)

PRIMARY OUTCOMES:
Core temperature | Up to 90 minutes
  Core temperature during exercise
Heart Rate | Up to 90 minutes
  Heart rate during exercise
Skin temperature | Up to 90 minutes
  Mean-weighted skin temperature during exercise
Whole-body sweat loss | 90 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin J Ryan, PhD, Principal Investigator — United States Army Research Institute of Environmental Medicine
Locations (1):
- US Army Research Institute of Environmental Medicine, Natick, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-04-26): https://cdn.clinicaltrials.gov/large-docs/53/NCT07080853/ICF_000.pdf